CLINICAL TRIAL: NCT07078812
Title: Comparison of Mirror Therapy and Action Observation Therapy on Upper Limb Sensory Motor Recovery and Quality of Life in Subacute Stroke Patients
Brief Title: Mirror Therapy and Action Observation Therapy on Upper Limb Sensory Motor Recovery and Quality of Life in Subacute Stroke Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lahore (Other)
Responsible Party: Principal Investigator, Komal Mushtaq, Student, University of Lahore
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UOL/IREB/25/09/0005
Record Dates: First submitted 2025-07-12; First posted 2025-07-22 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Stroke
Keywords: Action observation therapy; Mirror therapy; Quality of life; Stroke rehabilitation; Upper limb recovery
MeSH Terms: conditions — Stroke | interventions — Mirror Movement Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mirror Therapy for Upper Limb Rehabilitation (Experimental): Participants in this arm will undergo Mirror Therapy sessions targeting the affected upper limb. A mirror will be positioned along the patient's midline, reflecting movements of the non-paretic limb, creating the illusion of movement in the affected limb. Patients will perform bilateral symmetrical movements while observing the mirrored reflection for 30 minutes per session, 5 days per week, over a 6-week period. Standard stroke rehabilitation exercises will also be provided.
  Interventions: Behavioral: Mirror Therapy
- Action Observation Therapy for Upper Limb Rehabilitation (Experimental): Participants in this arm will receive Action Observation Therapy involving the observation of video clips demonstrating functional upper limb tasks, followed by physical practice of the same movements. Each session will consist of 15 minutes of video observation and 15 minutes of task execution, conducted 5 days per week for 6 weeks. This intervention will be supplemented by routine post-stroke rehabilitation exercises.
  Interventions: Behavioral: Action Observation Therapy

INTERVENTIONS:
Behavioral: Mirror Therapy — Mirror Therapy involves placing a mirror in the patient's midsagittal plane to reflect movements of the unaffected upper limb, creating a visual illusion of movement in the paretic limb. Patients perform bilateral symmetrical movements while focusing on the mirror reflection, helping to stimulate motor cortex activation and promote neuroplasticity. Sessions last 30 minutes, 5 days per week, for 6 weeks. This intervention is delivered in addition to standard stroke rehabilitation.
  Arms: Mirror Therapy for Upper Limb Rehabilitation
Behavioral: Action Observation Therapy — Action Observation Therapy consists of observing video demonstrations of functional upper limb movements, followed by the patient imitating the observed actions. Each session includes 15 minutes of watching goal-directed tasks and 15 minutes of active execution. This therapy aims to activate the mirror neuron system and enhance motor recovery. The protocol is administered 5 days per week for 6 weeks and is combined with routine stroke rehabilitation practices.
  Arms: Action Observation Therapy for Upper Limb Rehabilitation

SUMMARY:
This clinical study is being conducted to compare the effects of two different rehabilitation techniques-Mirror Therapy and Action Observation Therapy (AOT)-on improving upper limb movement and quality of life in individuals who have recently experienced a stroke. Stroke survivors often face weakness and coordination problems in their arms and hands. Helping them regain motor function is crucial for performing everyday tasks like dressing, eating, and writing.

Mirror Therapy works by having patients perform movements while watching the reflection of their unaffected limb in a mirror, tricking the brain into believing both limbs are working. This may help activate brain regions responsible for motor control.

Action Observation Therapy, on the other hand, involves patients watching videos of someone else performing arm and hand movements. After observing, patients try to mimic the actions themselves. This method is based on the theory that watching and imitating movements can enhance brain recovery.

In this study, patients will be randomly assigned to either the Mirror Therapy group or the Action Observation Therapy group. Both groups will receive therapy over several weeks, along with routine stroke rehabilitation care. Researchers will assess each patient's progress using standard tools to measure arm strength, hand coordination, and overall quality of life.

This study aims to find out which therapy leads to better recovery and could become a recommended part of post-stroke rehabilitation programs.

DETAILED DESCRIPTION:
Background Stroke is a major cause of adult disability worldwide. One of the most disabling consequences is upper limb impairment, which reduces independence and daily functioning. Although traditional rehabilitation helps, recovery is often incomplete. Therefore, innovative, neuroplasticity-driven therapies like Mirror Therapy (MT) and Action Observation Therapy (AOT) are gaining interest.

MT relies on visual feedback from a mirror to create an illusion of movement in the affected limb, activating motor cortical areas. AOT involves observing purposeful movement followed by imitation, leveraging the brain's mirror neuron system to promote recovery.

While both therapies have shown individual effectiveness, few studies have directly compared them in subacute stroke-a critical recovery window. This study aims to address that gap, offering evidence to inform clinical practice.

Objectives

Primary Objective:

To compare the effects of MT and AOT on upper limb sensorimotor recovery in individuals with subacute stroke.

Secondary Objective:

To assess the impact of these therapies on stroke survivors' quality of life.

Hypotheses

Null Hypothesis (H₀):

There is no significant difference between MT and AOT in improving motor function or quality of life.

Alternative Hypothesis (H₁):

There is a significant difference between the two interventions in enhancing motor recovery and life quality.

Study Design Type: Randomized Controlled Trial (RCT)

Setting: Outpatient Neurological Rehabilitation Center

Duration: 6-week intervention

Sample Size: 40 participants (20 per group)

Randomization: Block randomization with concealed allocation

Blinding: Assessor-blinded

Assessment Points: Baseline, Week 3, Week 6

Eligibility Criteria

Inclusion Criteria:

Aged 40-70 years

First-ever ischemic or hemorrhagic stroke (diagnosed via imaging)

Stroke onset within 6 months (subacute phase)

Hemiparesis involving upper limb

MMSE score ≥ 24

Medically stable

Exclusion Criteria:

MAS score > 2 (severe spasticity)

Cardiac instability or other severe comorbidities

Visual impairments affecting mirror or screen-based tasks

History of upper limb orthopedic surgeries

Enrolled in other rehabilitation trials

Intervention Groups Group A: Mirror Therapy (MT) Participants will perform upper limb tasks while viewing the mirrored reflection of their unaffected limb for 30 minutes/session, 5 days/week for 6 weeks.

Group B: Action Observation Therapy (AOT) Participants will observe upper limb task videos (15 min) followed by 15 minutes of physical practice of the same tasks, 5 days/week for 6 weeks.

All participants will continue to receive standard rehabilitation care, including physiotherapy and occupational therapy.

Outcome Measures

Primary Outcome:

Fugl-Meyer Assessment - Upper Extremity (FMA-UE):

Evaluates upper limb motor control and coordination.

Secondary Outcomes:

Stroke Impact Scale (SIS):

Assesses quality of life across physical and emotional domains.

Modified Ashworth Scale (MAS):

Quantifies muscle spasticity.

Box and Block Test:

Measures gross manual dexterity.

Motor Activity Log (MAL):

Evaluates the functional use of the affected arm in daily tasks.

Assessments will be conducted at three time points: baseline, week 3, and week 6.

ELIGIBILITY:
Inclusion Criteria:

* Age between 45 and 65 years (Tsai et al., 2012).
* Gender as either male or female (Tsai et al., 2012).
* Only subacute stroke patients will be included (Uyttenboogaart et al., 2005).
* A baseline Fugl-Meyer Assessment (FMA) score between 20 and 60 for upper limb motor function (Fugl-Meyer et al., 1975).
* The ability to follow study instructions, assessed using the Taiwan version of the Montreal Cognitive Assessment (MoCA) (Tsai et al., 2012), with scores below 26 indicating cognitive impairment, as patients scoring around 60 are considered to have near-normal cognitive function.
* The capability to participate in therapy and assessment sessions (Wang et al., 2011).
* Patient who have 1st onset of stroke ( 1st time stroke) (Hsieh et al., 2009).

Exclusion Criteria:

* Participants having hamonomus hemianopia (Tsai et al., 2012).
* Other neurological conditions for example, parkinsons, alzehmiers, ADHD, autism, etc (Tsai et al., 2012).
* Participants having recurrent stroke history (Wang et al., 2011).
* Global or receptive aphasia (Banks and Marotta, 2007).
* Severe neglect (Duncan et al., 2003).
* Major medical problems or comorbidities that influenced UE usage or cause severe pain (Hsieh et al., 2009).

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2024-11-15 (Actual); Primary Completion 2025-05-19 (Actual); Study Completion 2025-07-08 (Actual)

PRIMARY OUTCOMES:
Change in Upper Limb Motor Function as Measured by the Fugl-Meyer Assessment | Baseline, Week 3 (Mid-intervention), and Week 6 (Post-intervention)
  The Fugl-Meyer Assessment for Upper Extremity is a standardized, stroke-specific performance-based measure that evaluates motor functioning, balance, and joint coordination. The upper limb subscale (score range: 0-66) assesses voluntary movement, reflex activity, and coordination of the shoulder, elbow, forearm, wrist, and hand. A higher score indicates better motor function and recovery. This tool has strong psychometric properties and is widely used in stroke rehabilitation research to detect motor improvements over time.

SECONDARY OUTCOMES:
Change in Stroke-Related Disability (Modified Rankin Scale) | Baseline, Week 3, and Week 6
  The Modified Rankin Scale measures the degree of disability or dependence in daily activities following a stroke. It ranges from 0 (no symptoms) to 6 (death). Lower scores indicate better functional independence.
Change in Health-Related Quality of Life (Stroke Impact Scale - Version 3.0) | Baseline, Week 3, and Week 6
  The Stroke Impact Scale is a stroke-specific, self-reported questionnaire that assesses physical, emotional, and social aspects of recovery. It includes domains such as strength, mobility, memory, communication, and participation. Higher scores indicate better quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Lahore Teaching Hospital, Lahore, Pakistan

IPD SHARING:
Plan to Share IPD: No